CLINICAL TRIAL: NCT02211794
Title: A Prospective, Non-randomized, Consecutive Series, Multicenter, Observational Trial to Evaluate the Clinical Outcome of Total Knee Arthroplasty Using Journey II BCS Total Knee System
Brief Title: Journey II BCS EU Observational Trial
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: R11009-7
Record Dates: First submitted 2014-07-22; First posted 2014-08-07 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Degenerative Joint Disease
Keywords: Total Knee Arthroplasty; degenerative joint disease
MeSH Terms: conditions — Joint Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 cohort: subject requires primary total knee arthroplasty with the Journey II BCS Total Knee System, including patella resurfacing due to degenerative joint disease (primary osteoarthritis, post-traumatic arthritis, avascular necrosis, rheumatoid arthritis)
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection

SUMMARY:
Post-market study to confirm the safety and efficacy of the Journey II BCS knee prosthesis.

DETAILED DESCRIPTION:
Multicenter, prospective, observational study to collect relevant clinical data from 167 subjects implanted with the Journey II BCS Knee System. Data from eligible subjects, who have provided written informed consent for the collection of their coded data will be recorded from the patient's medical file on specially designed case report forms (CRF's).

Total study duration for participants will be 10 years with follow-up visits planned at 3 months, 1 year, 2 years, 5 years and 10 years post-surgery. An interim analysis describing the clinical outcome is planned after 5 years.

ELIGIBILITY:
Inclusion Criteria

* subject requires primary total knee arthroplasty with the Journey II BCS Total Knee System, including patella resurfacing
* subject requires primary total knee arthroplasty due to degenerative joint disease (primary osteoarthritis, post-traumatic arthritis, avascular necrosis, rheumatoid arthritis)
* subject is of legal age to consent, agrees to consent to and to follow the study visit schedule, by signing the EC approved informed consent form

Exclusion Criteria:

* age > 75 years
* conditions that may interfere with the TKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease)
* subject has inadequate bone stock to support the device

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a patient population consisting of 150 cases and recruited from 4 different countries, will be followed up when undergoing TKA as part of their standard care
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2014-01; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Revision for any reason | 10Years
  The goal of this study is to confirm the safety and efficacy of the Journey II BCS knee prosthesis by demonstrating non-inferiority of the cumulative percent success in subjects implanted with the JOURNEY II BCS Total Knee System compared to a literature reference rate of 94.3% (AOA annual report 201121) at 10 years. "Success" is defined as 10 year survival of the study device without revision for any reason.

SECONDARY OUTCOMES:
EQ-5D questionnaire | pre-op, 3month, 1yr, 2yr, 5yr, 10yr
  patient's opinion about his state of health, according to a visual analogue scale and 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression, (each dimension having 3 levels: no problems, some problems, extreme problems)
Knee Pain Evaluation Form questionnaire | 3month, 1yr, 2yr
  Assessment of post-operative knee pain
2011 Knee Society Score | pre-op, 3month, 1yr, 2yr, 5yr, 10yr
  A clinical follow-up and patient satisfaction, patient's expectations and a self-assessment of the physical outcome
radiographic evaluation | pre-op, discharge, 3month, 1yr, 5yr, 10yr
  The Knee Society Total Knee Arthroplasty Roentographic Evaluation and Scoring System will be used to analyse radiographic findings at each visit.
complication rate (adverse events and revisions) | discharge, 3month, 1yr, 2yr, 5yr, 10yr
  complications will be assessed at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Risebury, MD, Principal Investigator — North Hampshire Hospital; Fabio Catani, Prof, Study Chair — University of Modena and Reggio Emilia; Jan Victor, Prof, Principal Investigator — UZ Ghent; Gijs Van Hellemondt, Principal Investigator — Sint-Maartenskliniek Nijmegen; Stig Heir, Principal Investigator — Martina Hansens Hospital
Locations (5):
- UZ Gent, Ghent, Belgium
- University of Modena and Reggio Emilia, Modena, Italy
- Sint Maartenskliniek, Nijmegen, Netherlands
- Martina Hansens Hospital, Sandvika, Norway
- North Hampshire Hospital, Basingstoke, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
BSI Publication